CLINICAL TRIAL: NCT03650751
Title: Convenience Sampling，Clinical Study on Screening of Nursing Evaluation Indicators of Stroke Patients
Brief Title: Clinical Study on Screening of Nursing Evaluation Indicators of Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20173357201830
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: stroke；nursing assessment；condition of a patient；deterioration；
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stroke patients；neurologic impairment: It provides nursing staff with a unified reference standard for nursing observation indicators and sets monitoring and warning values according to the score, which is helpful to improve the timeliness and accuracy of nursing observation for patients with cerebral apoplexy.
  Interventions: Other: Nursing observation indexes

INTERVENTIONS:
Other: Nursing observation indexes — It provides nursing staff with a unified reference standard for nursing observation indicators and sets monitoring and warning values according to the score, which is helpful to improve the timeliness and accuracy of nursing observation for patients with cerebral apoplexy.

SUMMARY:
The purpose of this study was to use Delphi method to screen the nursing observation indexes of patients with stroke, and to screen the sensitive indexes with high correlation with the severity of stroke.It is used to guide nursing staff to observe the nursing of patients with cerebral apoplexy.

ELIGIBILITY:
Inclusion Criteria:

①according to the diagnostic criteria which was revisied in 1996 at the fourth national cerebrovascular disease conference,Patients were diagnosed with cerebral apoplexy through computerized tomographic scanning or Magnetic Resonance Imaging examination.

②Patients who volunteer to participate in the study and Sign the consent form.

Exclusion Criteria:

①Patients With other serious diseases, such as tumor, grade 2 or above of cardiac function.

②Had a history of mental illnes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Shenzhen 2nd People's Hospital ，Neurology wards
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
construct a nursing evaluation system for stroke patients | October 1st, 2017 - October 1st, 2018
  The nursing indexes of patients with cerebral apoplexy were selected. The nursing observation indexes of stroke patients were digitized and an electronic nursing evaluation sheet was formed.

CONTACTS AND LOCATIONS:
Overall Officials: xiaohua XIE, Master, Study Director — Shenzhen 2nd People's Hospital
Locations (1):
- Shenzhen second people's hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided